CLINICAL TRIAL: NCT04697784
Title: Post-Approval Study of the TREO Abdominal Stent-Graft System (P190015) in Patients With Infrarenal Abdominal Aortic and Aorto-iliac Aneurysms
Brief Title: Post-Approval Study of the TREO Abdominal Stent-Graft System
Acronym: TREO PAS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bolton Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IP-0021-20
Record Dates: First submitted 2020-12-10; First posted 2021-01-06 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: AAA; Abdominal Aortic Aneurysm; TREO; EVAR
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Intervention Model Description: Abdominal Aortic Aneurysm Stent-Graft
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Subjects who receive the TREO Abdominal Stent-Graft System (Experimental): Eligible subjects will be implanted with the TREO Abdominal Stent-Graft System.
  Interventions: Device: TREO Abdominal Stent-Graft System

INTERVENTIONS:
Device: TREO Abdominal Stent-Graft System — The TREO Abdominal Stent-Graft System is intended for the treatment of infrarenal abdominal aortic aneurysms with or without iliac involvement.

SUMMARY:
The purpose of this study is to determine the long-term performance of the TREO Abdominal Stent-Graft as a treatment for patients with Infrarenal Abdominal Aortic Aneurysms or Aorto-iliac Aneurysms.

DETAILED DESCRIPTION:
This is a prospective, multi-center, non-randomized, single-arm, post-market, non-interventional study of treatment with the TREO Abdominal Stent-Graft in subjects with Infrarenal Abdominal Aortic Aneurysms or Aorto-iliac Aneurysms. The study will include a minimum of 300 subjects treated with the TREO Abdominal Stent-Graft at up to 55 investigational sites in the US.

The primary objective is the collection of real world safety and effectiveness outcomes of the TREO Abdominal Stent-Graft System in an all-comers population eligible for the endovascular treatment of AAA in routine clinical practice, with emphasis on subjects that experience a device stent-strut or barb fracture.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to comply with all study procedures and visits.
* Written informed consent to participate in the study.
* Patient's aneurysm can be treated with the TREO Abdominal Stent-Graft System.
* Adequate data (medical records/imaging studies) available to analyze the primary endpoints for patients enrolled retrospectively.

Exclusion Criteria:

• Medical, social or psychological problems that, in the opinion of the investigator, preclude patient from receiving treatment with the TREO Abdominal Stent-Graft System.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of stent-strut fracture or barb separation as confirmed by the Imaging Core Laboratory. | Through 5 Years post-procedure
  Incidence of fracture in a stent-strut or separation of one or more proximal fixation barbs as confirmed by the Imaging Core Laboratory upon review of post-implant imaging studies.
Incidence of secondary intervention for adverse events related to or caused as a result of stent-strut fracture or barb separation. | Through 5 Years post-procedure
  Incidence of secondary intervention for adverse events related to or caused as a result of a fracture in a stent-strut or separation of one or more proximal fixation barbs. Relatedness to the device will be confirmed by the Clinical Events Committee (CEC) through review of available treatment and procedure records and reports of imaging studies.

SECONDARY OUTCOMES:
Number of participants with technical success at the conclusion of the index procedure | Through 5 Years post-procedure
  Defined as the following:
  * successful delivery (i.e., ability to deliver the implant to the intended location without the need for unanticipated corrective intervention related to delivery);
  * successful and accurate deployment (deployment of the endovascular stent graft in the planned location; patency of the endovascular stent graft, absence of device deformations such as kinks, stent eversion, mal-deployment, misaligned deployment, requiring unplanned placement of an additional device within the endovascular stent graft, and
  * successful withdrawal (i.e. successful withdrawal of the delivery system, without the need for unanticipated corrective intervention related to withdrawal)
Major Adverse Events | Through 5 Years post-procedure
  Incidence of the following Major Adverse Events
  * Myocardial infarction according to SCAI definition
  * Stroke according to the VARC-2 guidelines
  * New Onset Renal Failure requiring permanent dialysis
  * New onset Respiratory Failure requiring permanent home oxygen therapy through 30 days
  * Permanent Paralysis/Paraplegia
  * Bowel Ischemia
  * Procedural blood loss (≥ 1000cc)
Incidence of procedure-related clinical utility measures | Through 5 Years post-procedure
  Reporting of procedural data collected during implant of the TREO Abdominal Stent-Graft System including: Procedure time (minutes), Fluoroscopy time (minutes), Contrast volume (mL), Access method (i.e. percutaneous, surgical cut down), Length of ICU stay (hours), Length of hospital stay post-procedure (days), Anesthesia Type.
Incidence of procedure-related complications | Through 5 Years post-procedure
  Incidence of adverse events occurring during or following the implant determined by the CEC to be procedure-related.
Incidence of successful aneurysm treatment | 12 months post-implant
  Successful aneurysm treatment is defined as:
  * Technical success
  * Absence of death from the initial procedure, secondary intervention or aortic-related cause.
  * Absence of persistent type I or III endoleaks
  * Absence of aneurysm sac expansion >5 mm
  * Absence of device migration >10mm
  * Absence of failure due to device integrity issues
  * Absence of aneurysm rupture
  * Absence of conversion to open surgical repair
  * Absence of permanent paraplegia, disabling stroke or dialysis that resulted from the initial operation or a secondary intervention to treat the original aortic pathology.
Incidence of all-cause mortality | Through 5 Years post-procedure
  Rate of mortality attributed to any causality as confirmed by the CEC.
Incidence of aneurysm-related mortality | Through 5 Years post-procedure
  Rate of mortality attributed to the following causes as confirmed by the CEC: death due to a rupture, death within 30 days or prior to hospital discharge from primary procedure, or death within 30 days or prior to hospital discharge for a secondary procedure designed to treat the original aneurysm.
Incidence of aneurysm rupture | Through 5 Years post-procedure
  Incidence of rupture of the native aneurysm sac post-implantation of the endograft as confirmed by the CEC.
Incidence of secondary interventions. | Through 5 Years post-procedure
  Incidence of secondary procedures designed to treat or repair the original aneurysm treated with the TREO Abdominal Stent-Graft System
Incidence of conversion to open surgical repair. | Through 5 Years post-procedure
  Incidence of conversion to open surgical AAA repair during the initial EVAR procedure secondary to any procedure-related complications as determined by the CEC.
Incidence of stent-graft occlusion (i.e., loss of patency) | Through 5 Years post-procedure
  Incidence of stent-graft occlusion defined as the unintentional obstruction of the vascular/endograft lumen with minor obstruction (0-25%), minimal obstruction (26-74%), moderate obstruction (75-99%) or occlusion (100%) as confirmed by the Imaging Core Lab due to causes such as twisting or kinking of the prosthesis, oversizing and fabric pleating, or failure of the implant to fully open, or to mural thrombus deposition.
Incidence of device stenosis or kink | Through 5 Years post-procedure
  Incidence of stenosis or kinking of the TREO Stent-Graft as confirmed by the Imaging Core Lab.
Incidence of loss of device integrity | Through 5 Years post-procedure
  Incidence of changes in the structural integrity in a material component of the stent-graft such as a stent-strut fracture or separation of the proximal fixation barbs as confirmed by the Imaging Core Lab.
Incidence of aneurysm enlargement (>5mm as compared to 30-day imaging). | Through 5 Years post-procedure
  Incidence of the increase in the aneurysm sac diameter > 5 mm at post-implant follow-up visits relative to the diameter determined at the first post-procedural imaging study, as confirmed by the Imaging Core Lab.
Incidence of stent-graft migration (>10mm as compared to 30-day imaging) | Through 5 Years post-procedure
  Incidence of the longitudinal movement of all or part of a stent or attachment system for a distance of >10 mm relative to anatomical landmarks that were determined at the first post-procedural imaging study as confirmed by the Imaging Core Lab.
Incidence of Type I, II, III, IV or V Endoleaks | Through 5 Years post-procedure
  Incidence of Type I, II, III, IV or V Endoleaks defined as the persistence of blood flow outside the lumen of the stent-graft but within the native aorta or adjacent vascular segment being treated by the stent-graft as determined by the Imaging Core Lab.

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen Wild, Study Director — Terumo Aortic
Locations (40):
- United States (40):
  - Vascular Surgery Specialists, Phoenix, Arizona
  - Pima Heart and Vascular, Tucson, Arizona
  - University of California, San Francisco-Fresno, Fresno, California
  - University of California, San Diego, La Jolla, California
  - VA San Diego, San Diego, California
  - University of Colorado Anschutz, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Malcom Randall VA Medical Center, Gainesville, Florida
  - University of Florida, Gainesville, Florida
  - Coastal Vascular and Interventional, Pensacola, Florida
  - University of South Florida / Tampa General Hospital, Tampa, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - University of Iowa Hospital and Clinic, Iowa City, Iowa
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - McLaren Bay Region, Bay City, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Barnes Jewish Hospital at Washington University, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Rutgers Robert Wood Johnson Medical Center, New Brunswick, New Jersey
  - Lenox Hill Hospital / Northwell Health, New York, New York
  - Stony Brook Medical Center, Stony Brook, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - Mission Health, Asheville, North Carolina
  - East Carolina University, Greenville, North Carolina
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - VA Portland Healthcare System, Portland, Oregon
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Wellmont Cardiology Services, Kingsport, Tennessee
  - St. David's Healthcare (Cardiothoracic and Vascular Surgeons), Austin, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - Sentara Heart Hospital, Norfolk, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No